CLINICAL TRIAL: NCT00090363
Title: Randomized, Double-blind, Parallel-group, Placebo-controlled, Multi-centre Study to Assess ZD4054 (Zibotentan) in Pain-free or Mildly Symptomatic Patients With Prostate Cancer and Bone Metastases Who Have Rising Serum Prostate Specific Antigen (PSA)
Brief Title: ZD4054 (Zibotentan) in Pain-free or Mildly Symptomatic Patients With Prostate Cancer and Bone Metastases Who Have Rising Serum Prostate Specific Antigen (PSA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4320C00006; Trial 6; ZD4054; NCT00107146 (obsolete NCT alias)
Record Dates: First submitted 2004-08-25; First posted 2004-08-30 (Estimated); Results first posted 2012-09-03 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Prostate Cancer
Keywords: rising PSA; bone metastases; Clinical study; pain-free or mildly symptomatic
MeSH Terms: conditions — Prostatic Neoplasms | interventions — ZD4054

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Placebo (Placebo Comparator): Matching placebo oral tablet once daily, with best supportive care
  Interventions: Drug: Placebo
- ZD4054 10 mg (Experimental): ZD4054 10 mg oral tablet once daily, with best supportive care
  Interventions: Drug: ZD4054 10 mg
- ZD4054 15 mg (Experimental): ZD4054 15 mg oral tablet once daily, with best supportive care
  Interventions: Drug: ZD4054 15 mg

INTERVENTIONS:
Drug: ZD4054 15 mg — 15 mg oral tablet once daily
  Other Names: Zibotentan
  Arms: ZD4054 15 mg
Drug: Placebo
  Arms: Placebo
Drug: ZD4054 10 mg — 10mg oral tablet once daily
  Other Names: (Zibotentan)
  Arms: ZD4054 10 mg

SUMMARY:
This study is being carried out to see if ZD4054 (Zibotentan) is effective in treating prostate cancer and spread of cancer to the bone, and if so, how it compares with placebo (sugar pill). The study will also provide further information on the safety of ZD4054 (Zibotentan).

ELIGIBILITY:
Inclusion Criteria:

* Surgically or medically castrated
* Bone metastasis
* Rising PSA

Exclusion Criteria:

* Opiate use
* Prior chemotherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2004-07; Primary Completion 2008-12 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Emerging Oncology Medical Science Director, MD, Study Director — AstraZeneca
Locations (60):
- United States (7):
  - Research Site, Tucson, Arizona
  - Research Site, Los Angeles, California
  - Research Site, Gainsville, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Cleveland, Ohio
  - Research Site, Simpsonville, South Carolina
- Australia (4):
  - Research Site, Wolloongabba, Queensland
  - Research Site, Ashford, South Australia
  - Research Site, Wodonga, Victoria
  - Research Site, Nedlands
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Leuven
- Canada (5):
  - Research site, Vancouver, British Columbia
  - Research site, London, Ontario
  - Research site, Toronto, Ontario
  - Research site, Montreal, Quebec
  - Research site, Québec, Quebec
- Denmark (2):
  - Research Site, Aarhus
  - Research Site, Herlev
- Finland (5):
  - Research Site, Helsinki
  - Research Site, Joensuu
  - Research Site, OYS
  - Research Site, Seinäjoki
  - Research Site, Tampere
- France (5):
  - Research Site, Lille
  - Research Site, Montpellier
  - Research Site, Paris
  - Research site, Pontoise
  - Research Site, Toulouse
- Research Site, Jakarta, Indonesia
- Netherlands (6):
  - Research Site, Eindhoven
  - Research Site, Groningen
  - Research Site, Heerlen
  - Research Site, Leiden
  - Research Site, Rotterdam
  - Research Site, Utrecht
- Norway (7):
  - Research Site, Bergen
  - Research Site, Fredrikstad
  - Research Site, Moelv
  - Research Site, Oslo
  - Research Site, Tromsø
  - Research Site, Trondheim
  - Research Site, Tønsberg
- Poland (3):
  - Research Site, Bydgoszcz
  - Research Site, Katowice
  - Research Site, Warsaw
- Sweden (3):
  - Research Site, Gothenburg
  - Research Site, Malmo
  - Research Site, Stockholm
- Switzerland (2):
  - Research Site, Geneva
  - Research Site, Locarno
- United Kingdom (7):
  - Research Site, Birmingham
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Maidstone
  - Research Site, Manchester
  - Research Site, Newcastle
  - Research Site, York

REFERENCES:
- [Derived] James ND, Caty A, Borre M, Zonnenberg BA, Beuzeboc P, Morris T, Phung D, Dawson NA. Safety and efficacy of the specific endothelin-A receptor antagonist ZD4054 in patients with hormone-resistant prostate cancer and bone metastases who were pain free or mildly symptomatic: a double-blind, placebo-controlled, randomised, phase 2 trial. Eur Urol. 2009 May;55(5):1112-23. doi: 10.1016/j.eururo.2008.11.002. Epub 2008 Nov 29. PMID 19042080

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 447 patients with prostate cancer who had bone metastases with no pain or mild symptoms of pain and a rising serum Prostate Specific Antigen (PSA), despite a serum testosterone of <= 2.4 nmol/L (70 ng/dL), were recruited between 14th July 2004 and 10th January 2006.
Pre-assignment Details: 135 of the 447 enrolled patients were not randomised to treatments groups: 126 failed screening and 9 did not meet one or more of the study inclusion or exclusion criteria.
Period: Overall Study
Arm/Group | Placebo | ZD4054 10 mg | ZD4054 15 mg
Started | 107 | 107 | 98
Received Study Treatment. | 107 | 107 | 98
Completed | 1 (Number of patients receiving study treatment at data cut-off (18th December 2008).) | 0 (Number of patients receiving study treatment at data cut-off (18th December 2008).) | 2 (Number of patients receiving study treatment at data cut-off (18th December 2008).)
Not Completed | 106 | 107 | 96
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Withdrawal by Subject | 7 | 7 | 6
Not completed — Study-specific discontinuation criteria | 75 | 74 | 62
Not completed — Eligibility criteria not fulfilled | 0 | 0 | 1
Not completed — Consent expired | 7 | 10 | 9
Not completed — Reasons not specified | 2 | 1 | 1
Not completed — Continuing on study off treatment | 14 | 13 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ZD4054 10 mg | ZD4054 15 mg | Total
Number analyzed (Participants) | 107 | 107 | 98 | 312
Age Continuous [Mean (Standard Deviation); unit: years] | 71 (9) | 70 (8) | 69 (8) | 70 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 107 | 107 | 98 | 312
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 106 | 107 | 93 | 306
  Black | 0 | 0 | 1 | 1
  Oriental | 1 | 0 | 3 | 4
  Other | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic | 3 | 4 | 3 | 10
  African-American | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 3 | 4
  Japanese | 0 | 0 | 1 | 1
  Not a specific ethnic group | 99 | 95 | 87 | 281
  Other | 4 | 8 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (TTP)
Description: Median time (in days) from randomisation until disease progression, where progression is defined, using RECIST, as a measurable increase in the smallest dimension of any target or non-target lesion, or the appearance of new lesions, since baseline or death using the Kaplan-Meier method.
Time Frame: Follow-up for progression/death was 4-weekly for 2 years after first dose and 3-monthly thereafter. 'Final analysis' results are given - the most recent formal analysis (data cut-off 18th December 2008).
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo | ZD4054 10 mg | ZD4054 15 mg
Number analyzed (Participants) | 107 | 107 | 98
Days | 111 [77 to 252] | 138 [80 to 247] | 113 [80 to 279]

2. Secondary Outcome: Time to Death
Description: Median time (in days) from randomisation until death using the Kaplan-Meier method.
Time Frame: Follow-up for progression/death was 4-weekly for 2 years after first dose and 3-monthly thereafter. After progression survival was assessed 6-monthly. 'Final analysis' results are given - the most recent formal analysis (data cut-off 18th December 2008).
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo | ZD4054 10 mg | ZD4054 15 mg
Number analyzed (Participants) | 107 | 107 | 98
Days | 596 [317 to 893] | 706 [457 to 1043] | 717 [452 to 1232]

3. Secondary Outcome: Change in Total Prostate Specific Antigen (PSA) Over Time
Description: Percentage change in total Prostate Specific Antigen (PSA) (ng/mL) from baseline to 12 weeks.
Time Frame: Baseline to 12 weeks. 'Initial analysis' results are given - the most recent formal analysis (data cut-off 10th April 2006).
Population: The analysis population only includes patients with baseline and Week 12 PSA measurements
Measure: Mean (Standard Deviation); unit: Percentage Change in PSA
Arm/Group | Placebo | ZD4054 10 mg | ZD4054 15 mg
Number analyzed (Participants) | 63 | 69 | 56
Percentage Change in PSA | 110.4 (179.16) | 131.6 (454.35) | 69.34 (99.14)

4. Secondary Outcome: Objective Response Rate (ORR)
Description: Using the Response Evaluation Criteria in Solid Tumours (RECIST), an objective response (OR) is defined as a patient having a best overall response of either complete response (CR) or partial response (PR), which is subsequently confirmed as per RECIST. Objective Response Rate (ORR) is defined as the percentage of patients with OR.
Time Frame: For patients with measurable disease at baseline, Response Evaluation Criteria in Solid Tumours (RECIST) scans were 12-weekly from randomisation. 'Initial analysis' results are given - the most recent formal analysis (data cut-off 10th April 2006).
Population: Only patients with measurable disease at the baseline were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | ZD4054 10 mg | ZD4054 15 mg
Number analyzed (Participants) | 51 | 44 | 41
percentage of participants | 0 | 0 | 0

5. Secondary Outcome: Change in Number of Bone Metastases Over Time
Description: Percentage change in the number of bone metastases from baseline to last available post-baseline scan prior to discontinuation.
Time Frame: Baseline to last available post-baseline scan prior to discontinuation, up to maximum of 1164 days.
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Placebo | ZD4054 10 mg | ZD4054 15 mg
Number analyzed (Participants) | 107 | 107 | 98
Percentage Change | 187.1 (212.6) | 113.4 (195.6) | 189 (245.2)

ADVERSE EVENTS:
Arm/Group | Placebo | ZD4054 10 mg | ZD4054 15 mg
Serious Adverse Events (participants affected / at risk) | 26/107 | 18/107 | 16/98
Other Adverse Events (participants affected / at risk) | 93/107 | 86/107 | 87/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=107) | ZD4054 10 mg (N=107) | ZD4054 15 mg (N=98)
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 2
Left Ventricular Dysfunction (Cardiac disorders) | 1 | 1 | 0
Myocardial Ischaemia (Cardiac disorders) | 1 | 0 | 0
Cardiac Failure (Cardiac disorders) | 0 | 3 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1 | 0
Cardiopulmonary Failure (Cardiac disorders) | 0 | 2 | 0
Sick Sinus Syndrome (Cardiac disorders) | 0 | 1 | 0
Macular Hole (Eye disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Proctitis Haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Small Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 0
Feeling Hot (General disorders) | 1 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 1 | 0
Oedema Peripheral (General disorders) | 1 | 0 | 0
Catheter Related Complication (General disorders) | 0 | 0 | 1
Chest Discomfort (General disorders) | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Lung Infection (Infections and infestations) | 0 | 1 | 0
Neutropenic Sepsis (Infections and infestations) | 0 | 0 | 1
Pneumonia Bacterial (Infections and infestations) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Soft Tissue Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases To Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Benign Colonic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases To Lymph Nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Loss Of Consciousness (Nervous system disorders) | 1 | 0 | 0
Cerebral Haemorrhage (Nervous system disorders) | 0 | 0 | 1
Spinal Cord Compression (Nervous system disorders) | 0 | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 2
Bladder Neck Obstruction (Renal and urinary disorders) | 1 | 0 | 0
Bladder Obstruction (Renal and urinary disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 1 | 0 | 0
Calculus Bladder (Renal and urinary disorders) | 0 | 1 | 0
Pyelocaliectasis (Renal and urinary disorders) | 0 | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Aortic Aneurysm Rupture (Vascular disorders) | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=107) | ZD4054 10 mg (N=107) | ZD4054 15 mg (N=98)
Abdominal Pain (Gastrointestinal disorders) | 6 | 0 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 7 | 0 | 3
Anaemia (Blood and lymphatic system disorders) | 7 | 6 | 3
Anorexia (Metabolism and nutrition disorders) | 10 | 12 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 10 | 8
Back Pain (Musculoskeletal and connective tissue disorders) | 19 | 18 | 17
Bone Pain (Musculoskeletal and connective tissue disorders) | 6 | 10 | 8
Constipation (Gastrointestinal disorders) | 11 | 13 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 7
Depression (Psychiatric disorders) | 1 | 6 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 7 | 7
Dizziness (Nervous system disorders) | 3 | 8 | 8
Dry Mouth (Gastrointestinal disorders) | 9 | 7 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 17 | 6
Fatigue (General disorders) | 7 | 18 | 10
Flushing (Vascular disorders) | 6 | 5 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 7
Haematuria (Renal and urinary disorders) | 4 | 6 | 4
Headache (Nervous system disorders) | 44 | 39 | 13
Hot Flush (Vascular disorders) | 8 | 5 | 6
Influenza (Infections and infestations) | 4 | 6 | 5
Insomnia (Psychiatric disorders) | 11 | 6 | 10
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 6
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 8 | 4 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 6 | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 34 | 31 | 4
Nasopharyngitis (Infections and infestations) | 8 | 5 | 8
Nausea (Gastrointestinal disorders) | 13 | 19 | 20
Oedema Peripheral (General disorders) | 47 | 42 | 11
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 7 | 10 | 12
Pollakiuria (Renal and urinary disorders) | 1 | 7 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 5
Pyrexia (General disorders) | 7 | 5 | 5
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 15 | 17 | 3
Urinary Tract Infection (Infections and infestations) | 3 | 3 | 8
Vomiting (Gastrointestinal disorders) | 7 | 6 | 9

LIMITATIONS AND CAVEATS:
'Final analysis' results (data cut-off 18th December 2008) should be considered in context with the longevity of the follow-up (median duration approximately 22 months) relative to only approximately 4 months median duration of study treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AstraZeneca can review results communications prior to public release and may within 30 days of receipt require that submission or disclosure be delayed for up to 2 months in order to file patent applications. AstraZeneca can also, within 30 days of receipt, require amendments to be made in order to protect its patent and / or corporate interests.